CLINICAL TRIAL: NCT01729741
Title: Drain or no Drain After Thyroid Surgery: a Randomized Clinical Trial at Mulago Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Department of Surgery (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Rec Ref 2010-139
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2010-12

CONDITIONS: Hospital Admission Duration; Postoperative Hematoma Formation; Wound Sepsis
Keywords: Drain or no drain; Thyroid surgery; Randomized Trial
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No drain (No Intervention): No drain was inserted after Thyroid surgery
- Drain (Experimental): A drain was inserted after thyroid surgery
  Interventions: Procedure: drain was inserted after thyroid surgery

INTERVENTIONS:
Procedure: drain was inserted after thyroid surgery — insertion of drain after thyroid surgery
  Other Names: drains; thyroid surgery
  Arms: Drain

SUMMARY:
Thyroidectomy is one of the most commonly performed operations in general surgery. Available data seem to suggest an association between no-drain usage and a shorter duration of hospital stay. Seung et al found that the (following thyroidectomy) time to discharge after thyroidectomy was significantly shorter in the no drain group compared to the drain group. Similar results were recorded in a study conducted by Davari et al. Hyoung et al reported the incidence of hematoma formation post- thyroidectomy to be varying between 0.3%-4.3%. Tahsin et al reported that post-thyroidectomy bleeding is as rare as 0.3%-1.0%. The fear of an hematoma enlarging and obstructing the airway and causing difficulty in breathing, prompts many surgeons to use drains routinely after any type of thyroid surgery. The main reason is to drain off a possible postoperative hemorrhage, which may compress the airway and produce respiratory fail

DETAILED DESCRIPTION:
This study will be aimed at comparing the patient outcomes with drain and no-drain insertion methods after thyroidectomy in a resource limited setting.

Study population: All adult patients aged between 18 to 79 years who attended the endocrinology outpatient clinic and had been diagnosed with goiter.

Study Participants: All adult patients with goiters who were eligible for thyroidectomy Inclusion criteria: All adult patients aged between 18 to 79 years with a diagnosis of goiter who consented to participate in the study.

Exclusion criteria: The investigators excluded patients with goiter who had a history suggestive of bleeding tendencies, recurrent goiter, and thyroid cancer with fixation of the thyroid gland to surrounding structures and had uncontrolled co-morbidities such as diabetes mellitus (DM) and hypertension (HT).

Inserting a drain after goiter surgery and not inserting a drain is the intervention all participants receive the same treatment

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged between 18 to 79 years with a diagnosis of goiter who consented to participate in the study

Exclusion Criteria:

* We excluded patients with goiter who had a history suggestive of bleeding tendencies, recurrent goiter, and thyroid cancer with fixation of the thyroid gland to surrounding structures and had uncontrolled co-morbidities such as diabetes mellitus (DM) and hypertension (HT).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay | 7 days
  Duration of hospital stay

SECONDARY OUTCOMES:
Haematoma formation | 7 days
  post operative complication

OTHER OUTCOMES:
wound sepsis | 7 days
  post operative wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Jane O Fualal, MD, Study Chair — Mulago Hospital, Uganda
Locations (2):
- Uganda (2):
  - Makerere University, Kampala
  - Mulago Hospital, Kampala

REFERENCES:
- [Background] Khanna J, Mohil RS, Chintamani, Bhatnagar D, Mittal MK, Sahoo M, Mehrotra M. Is the routine drainage after surgery for thyroid necessary? A prospective randomized clinical study [ISRCTN63623153]. BMC Surg. 2005 May 19;5:11. doi: 10.1186/1471-2482-5-11. PMID 15946379